CLINICAL TRIAL: NCT06084611
Title: Long Term Effects of Heat and Moisture Exchangers (HMEs) (Provox® Life™) on Pulmonary Symptoms in Laryngectomized Patients
Brief Title: Long Term Effects of Heat and Moisture Exchangers (HMEs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Collaborators: Instituto de Cancer Dr Arnaldo (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL_Brazil
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Laryngectomy; Status
Keywords: Laryngectomy; Heat and Moisture Exchanger; HME; Pulmonary rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Provox Life HME (Experimental): Use of Provox Life HMEs and attachment
  Interventions: Device: Provox Life
- Control - No HME (No Intervention): Control group is current standard of Care in Brazil, which is not using an HME

INTERVENTIONS:
Device: Provox Life — Compliant use of Provox Life HMEs
  Arms: Provox Life HME

SUMMARY:
Assessment of long term effect of Provox Life HME use on pulmonary symptoms in laryngectomized patients.

ELIGIBILITY:
Inclusion Criteria:

* Total laryngectomy, irrespective of pharynx reconstruction method
* 18 years or older
* Longer than 3 months after total laryngectomy
* Longer than 6 weeks after postoperative radiotherapy

Exclusion Criteria:

* Current use of HMEs (within last 3 months)
* Medical problems prohibiting the use of HME
* Active recurrent or metastatic disease (medical deterioration)
* Recent pulmonary infections/unstable pulmonary condition
* Insufficient physical, cognitive, or mental ability required to attach, remove or operate the devices themselves
* Low tidal volumes
* Unable to understand the Participant Information and/or unable to give Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
CASA-Q Score | Baseline, 3 months, 6 months, 9 months
  assessed with validated Coughing and Sputum Assessment Questionnaire (CASA-Q). Score between 0 and 100, with higher scores meaning less symptoms and less impact.

SECONDARY OUTCOMES:
Number of involuntary coughs per 24 hours | Baseline, 3 months, 6 months, 9 months
  Patient reported, recorded by tally sheeting
Forced Expectoration | Baseline, 3 months, 6 months, 9 months
  Patient reported, recorded by tally sheeting
Quality of Life by EQ-5D-5L | Baseline, 3 months, 6 months, 9 months
  patient reported, the descriptive system assesses health in five dimensions, from which a health state index score is calculated, range from 0 to 1, with higher scores indicating higher health utility
Jenkins sleep evaluation questionnaire | Baseline, 3 months, 6 months, 9 months
  Patient reported to assess sleep quality. Score between 0 and 20, with higher score the more sleep disturbances
Questionnaire to assess Shortness of Breath | Baseline, 3 months, 6 months, 9 months
  from Ackerstaff et al., 1993
Voice handicap Index | Baseline, 3 months, 6 months, 9 months
  patient reported outcome, score from 0-40, with higher scores indicating greater voice-related handicap.
Consumption of medical devices (Number of devices used) | Baseline, 3 months, 6 months, 9 months
  Number of devices used, by use of patient diary recoding number of devices used
Study-specific questionnaire to assess number of complications and medical treatments | Baseline, 3 months, 6 months, 9 months
  Study specific questionnaire to record complications and consumption of medications, diagnostics, treatment, medical care, medical transportation, sick leave

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cancer Dr. Arnaldo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No